CLINICAL TRIAL: NCT07048314
Title: A Randomized Clinical Trial to Assess Safety and Efficacy of Allogeneic Adipose-derived Mesenchymal Stem Cells in Promoting the Recovery of Erectile Function Post Radical Retropubic Prostatectomy of Localized Prostate Cancer
Brief Title: Stem Cells for Erectile Dysfunction Post RALP
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Brian Miles, MD, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00039638
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Erectile Dysfunction; Prostate Cancer
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms | interventions — Saline Solution; Ambulatory Care Facilities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1: allogeneic adipose-derived mesnchymal stem cells plus saline solution (Experimental): 2.00x 10⁸ HB-adMSCCs locally injected into the corpora cavernosa of the penis and along the right and left neurovascular bundle of the penis in the OR at week 1 plus Placebo via IV in clinic at week 12.
  Interventions: Drug: Allogeneic adipose-derived mesenchymal stem cells (HB-adMSCs) in the OR; Drug: Placebo in clinic
- 2: Placebo plus allogeneic adipose-derived mesnchymal stem cells (Experimental): 4 cc of saline solution in the corpora cavernosa of the penis and 4 cc of saline solution along the right and left neurovascular bundles of the penis in the OR at week 1 plus 2.00x 10⁸ HB-adMSCs via IV in clinic at week 12.
  Interventions: Drug: Allogeneic adipose-derived mesenchymal stem cells (HB-adMSCs) at the doctor's office; Drug: Placebo in the OR
- 3: allogeneic adipose-derived mesnchymal stem cells intra op and at week 12 in clinic (Experimental): 2.00x 10⁸ HB-adMSCs locally injected into the corpora cavernosa of the penis and along the right and left neurovascular bundle of the penis in the OR at week 1 plus 2.00x 10⁸ HB-adMSCs via IV in clinic at week 12.
  Interventions: Drug: Allogeneic adipose-derived mesenchymal stem cells (HB-adMSCs) at the doctor's office; Drug: Allogeneic adipose-derived mesenchymal stem cells (HB-adMSCs) in the OR
- 4: placebo plus placebo (Placebo Comparator): 4 cc of saline solution in the corpora cavernosa of the penis and 4 cc of saline solution along the right and left neurovascular bundles of the penis in the OR at week 1 plus saline solutin via IV in clinic at week 12.
  Interventions: Drug: Placebo in the OR; Drug: Placebo in clinic

INTERVENTIONS:
Drug: Allogeneic adipose-derived mesenchymal stem cells (HB-adMSCs) at the doctor's office — 2.00x10⁸ HB-adMSCs IV at the doctor's office.
  Other Names: HB-adMSCs
  Arms: 2: Placebo plus allogeneic adipose-derived mesnchymal stem cells; 3: allogeneic adipose-derived mesnchymal stem cells intra op and at week 12 in clinic
Drug: Allogeneic adipose-derived mesenchymal stem cells (HB-adMSCs) in the OR — 100 million stem cells (1.00x10⁸ HB-adMSCs) in the corpora cavernosa of the penis suspended in a 4 cc of sterile saline. 50 million stem cells (5.0x 10⁷ HB-adMSCs) along the right neurovascular bundle and 50 million cell (5.0x 10⁷ HB-adMSCs) along the left neurovascular bundle of the penis suspended in a 4 cc of sterile saline during the surgery
  Other Names: HB-adMSCs
  Arms: 1: allogeneic adipose-derived mesnchymal stem cells plus saline solution; 3: allogeneic adipose-derived mesnchymal stem cells intra op and at week 12 in clinic
Drug: Placebo in the OR — 4 cc of saline solution in the corpora cavernosa of the penis and 4 cc of saline solution along the right and left neurovascular bundles of the penis during the surgery .
  Other Names: Saline solution in the OR
  Arms: 2: Placebo plus allogeneic adipose-derived mesnchymal stem cells; 4: placebo plus placebo
Drug: Placebo in clinic — 30 mL syringe of the product should be mixed into a 250cc bag of sodium chloride solution 0.9% for infusion. should be administered intravenously, with a dosing rate of 4-5mL/min.
  Other Names: Saline solution in clinic
  Arms: 1: allogeneic adipose-derived mesnchymal stem cells plus saline solution; 4: placebo plus placebo

SUMMARY:
This is a phase 1/2 single center, pilot study to assess safety and efficacy of allogeneic adipose-derived mesenchymal stem cells (HB-adMSCs) and to evaluate the timing and combination effects of active treatment versus placebo in promoting the recovery of erectile function in patients undergoing radical retropubic prostatectomy (RALP) of localized prostate cancer.

DETAILED DESCRIPTION:
This is a prospective, single-center, double blind, four-arm, pilot study to evaluate safety and effectiveness of allogeneic stem cells promoting the recovery of erectile function in patients undergoing radical retropubic prostatectomy (RALP) of localized prostate cancer.

All participants will be assessed for eligibility Participants will be randomized in a 1:1:1:1 ratio to Arm 1, Arm 2, Arm 3 or Arm 4 using a validated system that automates the random assignment of participant numbers to randomization numbers.

Study participants will be randomized to receive either:

Arm 1 2.00x 10⁸ HB-adMSCCs locally injected into the corpora cavernosa of the penis and along the right and left neurovascular bundle of the penis in the OR at week 1 plus Placebo via IV in clinic at week 12.

Arm 2 Placebo locally injected into the corpora cavernosa of the penis and along the right and left neurovascular bundle of the penis in the OR at week 1 plus 2.00x 10⁸ HB-adMSCs via IV in clinic at week 12.

Arm 3 2.00x 10⁸ HB-adMSCs locally injected into the corpora cavernosa of the penis and along the right and left neurovascular bundle of the penis in the OR at week 1 plus 2.00x 10⁸ HB-adMSCs via IV in clinic at week 12.

Arm 4 Placebo locally injected into the corpora cavernosa of the penis and along the right and left neurovascular bundle of the penis in the OR at week 1 plus Placebo via IV in clinic at week 12.

Study Medication:

1. Stem cells locally injected in the penis: subjects will receive 1.00x 10⁸ HB-adMSCs injection into the corpora cavernosa of the penis and 5.0x10⁷ HB-adMSCs along the right neurovascular bundle and 5.0x10⁷ HB-adMSCs along the left neurovascular bundle during surgery in the Operating Room (OR)
2. Stem cells delivered intravenous: Subject will receive 2.00x10⁸ HB-adMSCs IV at the doctor's office.

The treatment duration will be 2 cycles. Treatment will be administered on Week 1 (in the OR) and on week 12 in the Urology Clinic.

The study duration will be 24 weeks post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for RALP with Dr. B. Miles at Houston Methodist.
2. Men aged between 40 and 70 (inclusive) years old
3. Localized prostate cancer: Clinical stage T1-T2, N0, M0
4. Gleason score < 7
5. Pre-op IIEF-5 >20 (Appendix A)
6. Testosterone serum: > 300ng/dl with normal Free Testosterone
7. Life expectancy of at least 10 years
8. Performance status of ≤ 2 (Zubrod scale). (Appendix B)
9. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with the policies of the institution
10. Patient is willing to attempt intercourse at least 5 times per month following urinary control after surgery
11. Supportive partner willing to complete sexual survey questionnaire (Appendix D)
12. PDE5 inhibitors like sildenafil, tadalafil, vardenafil and avanafil are permitted pre and post-surgery if participant was taking this for ED at least 6 months before surgery.
13. Patient need cardiac clearance by the cardiologist

Exclusion Criteria:

1. Penile anatomical abnormalities (Peyronie's disease)
2. Hypogonadism
3. Any medication used for androgen ablation (e.g., LHRH agonist or antagonist, anti-androgens, etc.)
4. Patients with AST levels above 40U/L ; ALT levels above 33 U/L and Glucose levels above 180 mg/dl and psychiatric disorders that require medication
5. Previous or current hormonal treatment, chemotherapy, radiation therapy, immunotherapy or another investigational drug.
6. Any previous penile implant or penile vascular surgery
7. Injections of Trimix (combination of alprostadil, papaverine and phentolamine) pre and post-surgery .

   -

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in erectile function by IIEF | from baseline to 6 months post treatment
  IIEF-5 is a tool to asses erectile dysfunction base on five questions about confidence, hardness, maintenance and satisfaction of erections. Score: 1 to 25.
Change in erectile function by Epic 26 | from baseline to 6 months post treatment
  This questionnaire is designated to measure Quality of Life issues.Clinical relevance (>12 points) for sexual function domain score as measured by EPIC-26.
Number of Participants With Severe Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-Related AEs, Deaths, Discontinuation of Study Drug Due to AEs, Immune-Related Adverse Events (irAE) | 6 months
  AE=any new unfavorable symptom, sign or disease or worsening of a preexisting condition that may not have a causal relationship with treatment.
  SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity or drug dependency/abuse; is life-threatening, an important medical event or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible or missing relationship to study drug. Death=during study and up to 70 days after last dose. IrAEs=AEs potentially associated with inflammation and considered to be causally related to study drug

SECONDARY OUTCOMES:
Change in urinary function | from baseline to 6 months post treatment
  This questionnaire is designated to measure Quality of Life issues.Clinically relevant (≥9 points) difference in the EPIC-26 urinary incontinence domain score

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist, Houston, Texas, United States